CLINICAL TRIAL: NCT05099250
Title: Evaluation of the Efficacy of Adding Magnesium Sulfate as an Adjuvant to Bupivacaine in Bilateral Ultrasound Guided Paravertebral Block for Laparoscopic Cholecystectomy
Brief Title: Adding Magnesium Sulfate to Bupivacaine in Ultrasound Guided Paravertebral Block for Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Marwa Ibrahim Mohamed Abdo,MD, Lecturer of Anesthesia and Surgical Intensive Care-Faculty of Medicine - Mansoura University, Mansoura University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS/18.01.12
Record Dates: First submitted 2021-08-19; First posted 2021-10-29 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: paravertebral block laparoscopic cholecystectomy
MeSH Terms: interventions — Bupivacaine; Sodium Chloride; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: The groups allocated are concealed in sealed opaque envelopes which were not opened until patient consent was obtained.
  The two groups were:
  1. Control group: Bupivacaine Group (B group) N=25 :
     Included patients who received 17 mL of 0.25% bupivacaine + 3 mL saline 0.9% in a total volume of 20 ml on each side.
  2. Magnesium Group (M group) N=25 :
  Included patients who received 17 mL of 0.25% bupivacaine + 3 mL of 75 mg magnesium sulfate diluted in 0.9% saline in a total volume of 20 ml on each side.
  All patients were performed by the same anesthetic team with standard procedure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The groups allocated are concealed in sealed opaque envelopes which were not opened until patient consent was obtained.
  The two groups were:
  1. Control group: Bupivacaine Group (B group) N=25 :
     Included patients who received 17 mL of 0.25% bupivacaine + 3 mL saline 0.9% in a total volume of 20 ml on each side.
  2. Magnesium Group (M group) N=25 :
  Included patients who received 17 mL of 0.25% bupivacaine + 3 mL of 75 mg magnesium sulfate diluted in 0.9% saline in a total volume of 20 ml on each side.
  All patients were performed by the same anesthetic team with standard procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: Bupivacaine Group (B group) (Placebo Comparator): Included patients who received 17 mL of 0.25% bupivacaine + 3 mL saline 0.9% in a total volume of 20 ml on each side
  Interventions: Drug: Bupivacain; Other: saline
- Magnesium Group (M group) (Active Comparator): Included patients who received 17 mL of 0.25% bupivacaine + 3 mL of 75 mg magnesium sulfate diluted in 0.9% saline in a total volume of 20 ml on each side.
  Interventions: Drug: Bupivacain; Drug: magnesium sulfate; Other: saline

INTERVENTIONS:
Drug: Bupivacain — local anesthetic agent
  Other Names: Control group: Bupivacaine Group (B group; Saline
Drug: magnesium sulfate — In the central nervous system , it has depressant effects, by antagonism at NMDA receptors and through inhibition of release of catecholamines
  Other Names: Magnesium Group (M group); saline
  Arms: Magnesium Group (M group)
Other: saline — medical solution

SUMMARY:
Laparoscopic cholecystectomy is one of the most commonly performed minimally invasive surgical procedures for the treatment of symptomatic cholelithiasis Laparoscopic cholecystectomy has clear benefits when compared with open surgery, but post-operative pain is still a common complaint after it The patient undergoing laparoscopic cholecystectomy suffers from severe post-operative pain, it can prolong hospital stay and lead to increased morbidity Post-operative laparoscopic cholecystectomy pain can be relieved by some methods pre-emptive analgesic regimens containing ketamine, regional anesthesia techniques including paravertebral block Paravertebral Block is a regional anesthetic and analgesic technique which may offer comparable analgesic effectiveness with minimal side effects Paravertebral Block has been used a lot in the last two decades, several studies show its efficacy in, thoracoscopic surgery and laparoscopic cholecystectomy .Paravertebral block is the technique of injecting local anesthetic adjacent to the thoracic vertebra close to where the spinal nerves emerge from the intervertebral foramina, resulting in ipsilateral somatic and sympathetic nerve blockade in multiple dermatomes above and below the site of injection .

Bupivacaine is a local anesthetic that is capable of producing prolonged high quality analgesia in the postoperative period It is shown that paravertebral block using bupivacaine significantly reduces pain score Many drugs have been used as adjuvants to local anesthetic in peripheral nerve block in order to augment its analgesic effect and prolong the duration of the block such as opioids and magnesium sulfate Many studies have reported safety and efficacy of adding magnesium to local anesthetics in various regional anesthetic procedures, such as intrathecal, epidural, caudal, brachial plexus blocks and intravenous regional anesthesia. Magnesium play a major role in central nociceptive transmission, modulation and sensitization of acute and chronic pain states due to its antagonistic effect on N-methyl D-aspartate (NMDA) receptors .

DETAILED DESCRIPTION:
Patients and Methods

Patients:

This is a blind prospective randomized controlled study that will be conducted for one year in Mansoura university hospitals after approval from the Institutional Research Board (IRB), Faculty of Medicine, Mansoura University, patients will be interviewed and written informed consents will be obtained. This study will include 26 patients of American Society of Anesthesiologists physical status grade I and grade II, of both sexes, aged between 20-60 years who will be scheduled for laparoscopic cholecystectomy.

Sample size calculation A Priori G-power analysis was done to estimate study sample size. A power of 90% was estimated with type I error of 0.05 to get an analgesic duration difference between groups of approximately 30% to yield of total sample size of 50 cases (25cases per group).

Randomization:

Fifty patients (number = 50) had laparoscopic cholecystectomy and bilateral paravertebral block during the study period. These patients were randomly allocated to undergo bilateral ultrasound guided paravertebral block. The groups allocated are concealed in sealed opaque envelopes which were not opened until patient consent was obtained.

The two groups were:

1. Control group: Bupivacaine Group (B group) Number=25 :

   Included patients who received 17 mL of 0.25% bupivacaine + 3 mL mili saline 0.9% in a total volume of 20 ml on each side.
2. Magnesium Group (M group) N=25 :

Included patients who received 17 mL of 0.25% bupivacaine + 3 mL of 75 mg milgram magnesium sulfate diluted in 0.9% saline in a total volume of 20 ml on each side.

All patients were performed by the same anesthetic team with standard procedure.

Methodology:

Anesthetic Management:

Preoperative Management:

All patients will be visited a day prior to surgery and will be assessed preoperatively by History, physical examination and laboratory evaluation (complete blood picture, coagulation profile, liver function and renal function tests). The study protocol and paravertebral block procedure will be explained to all patients. All patients will be familiar with the use of 0-10 visual analogue scale score identifying 0 as no pain and 10 as worst imaginable pain. Patient fast 6-8 hour before the time of surgery.

On arrival of the patient to the operating room routine monitoring will be applied, peripheral intravenous cannula 20 gauge will be inserted and 0.9% saline will be started to be infused. All patients will be premedicated using midazolam 0.03 mg/kg kilo intravenous.

Paravertebral block will be performed before induction of general anesthesia.

Technique of ultrasound guided paravertebral nerve block:

* Standard precautions for the performance of ultrasound-guided nerve blocks will be followed which include continuous routine monitoring, the skin overlying the injection site should be free of signs of infection and prepped with an antiseptic solution.
* Patient will lay in the lateral position, paravertebral block will be done using a 38 mm mile meter broadband linear array ultrasound probe.The probe surface in contact with the skin should be covered with a sterile adhesive dressing.
* A sagittal paramedian view of the paravertebral space will be obtained by applying the probe at a point 2.5 cm centimeter lateral to the tip of the spinous process in a vertical orientation, The fifth thoracic vertebral level will be identified by palpating and counting down from the seventh cervical body.
* The midpoint of the transducer will be aligned midway between the transverse processes of thoracic vertebra T5 and T6, 4 ml of 1 % lidocaine was injected subcutaneously at the puncture site,and 22 gauge spinal needle will be inserted in an in plane approach in a cephalad orientation and will be advanced perpendicularly to all skin planes under direct vision to puncture the superior costotransverse ligament where a click may be appreciated.
* Following negative aspiration, 1-2 ml of study solution will be injected to verify correct position of the needle tip and the rest of study solution will be injected in fractioned doses following intermittent aspiration between the superior costotransverse ligament and the parietal pleura which will be displaced anteriorly by the injectate.
* Similar approach will be used for the paravertebral block on the other side.
* Sensory block over the area of surgical incision will be confirmed by loss of cold sensation using an alcohol swab and pinprick sensation using a 23 G gauge needle every 3 mint until 15 min after injection of the study solutions and before starting general anesthesia.

General Anesthesia:

General Anesthesia will be induced using intravenous propofol (2-3 mg/kg), fentanyl IV (1µ/kg) microgram/kilo and atracurium besylate (0.6 mg/kg) to facilitate intubation. Then patient will be mechanically ventilated using a volume control mode with Tv 6-8ml/kg, respiratory rate 10-14 breath/min and I.E. ratio 1:2 to maintain Etco2 35-40 mmHg mli mercury. Anesthesia will be maintained using minimum alveolar concentration of isoflurane 1.2% and 60% air in O2 mixture with top up dose of atracurium. Intraoperative IV fluids will be given per body weight and according to intraoperative loss.

All patients will be extubated at the end of surgery after neuromuscular reversal with administration of neostigmine (0.05 mg/kg) and IV atropine (0.02 mg/kg) and fulfilling the criteria of extubation. The duration of the surgery will be recorded.

Monitoring:

Intra-operative assessment

* In operating room, monitoring will be achieved by five lead electro cardi gram, oxygen saturation and non-invasive mean arterial blood pressure.
* Base line values of heart rate, oxygen saturation and non-invasive mean arterial blood pressure will be collected before and after paravertebral block, just after induction of anesthesia, at skin incision, then recording will be done every 15 mint till the end of the first hour and then every 30min interval till the end of surgery.
* Sensory block onset will be defined when the patient subjectively evaluate the intensities of both cold and pinprick sensations in the blocked side decrease 75 % or more.
* Duration of surgery will be defined as the time from induction to discharge from the operating room will be recorded.
* In case of increased in intra-operative systolic blood pressure and heart rate of more than 20% of baseline for longer than 5min, incremental doses of fentanyl IV 0.5µ/kg will be given and the case will be excluded.

Postoperative Assessment:

* On admission into the post operative care unit, all vital data & hemodynamics (non-invasive mean arterial blood pressure, heart rate, and oxygen saturation) will be recorded at 1, 2, 6, 12 and 24 hrs. postoperative
* Post-operative complications will be recorded including post-operative nausea and vomiting treated by metoclopramide, hypotension treated by phenylephrine drops, bradycardia treated by atropine or pneumothorax, respiratory depression and chest pain, respiratory depression is defined as respiratory rate less than 8 per minute or oxygen saturation below 90%.

Statistical analysis The statistical analysis of data will be done by using excel program for figures and Statistical Package for Social Science program version 22. To test the normality of data distribution Kolmogorov- Smirnov test will be done only significant data revealed to be nonparametric. Unpaired student-t test will be used for comparisons of numerical variables between-group, if its assumptions were fulfilled, otherwise for non-parametric; the Mann-Whitney test will be used. The description of data done in the form of mean (±SD) stander division for quantitative data and frequency and proportion for qualitative data. Any difference or change showing probability (P) less than 0.05 will be considered statistically significant at confidence interval 95%.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective laparoscopic cholecystectomy were enrolled in this study

Exclusion Criteria:

* patient refusal to participate,
* Sever renal or cardiac illness,
* Pulmonary diseases as emphysema or chronic obstructive pulmonary disease
* Neuromuscular diseases (as myopathies and myasthenia gravies), -Hematological diseases, bleeding or coagulation abnormality,
* Psychiatric diseases,
* Local skin infection and sepsis at site of the block,
* Known hypersensitivity to the study drugs, and Severe chest wall deformity, e.g. scoliosis.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
change of postoperative pain intensity | first 24 hours postoperatively
  measured by visual analogue scale . All patients were familiar with the use of 0 -10 visual analogue scale identifying 0 as no pain and 10 as worst imaginable pain.
  Pain intensity was assessed at rest and during cough with VAS score at 1, 2, 6, 12 and 24 hours postoperatively.
  When the patients experienced pain (VAS score > 3), A bolus dose of IV morphine 0.02 mg/kg was administered till visual analogue scale score ≤ 4 was attained.

SECONDARY OUTCOMES:
change opioid consumption in first 24 hours | first 24 hours postoperatively
  measured by recording the time of first post-operative administration of morphine.
  Also, the total dose of post-operative morphine (mg) consumed in the first postoperative 24 hours was calculated in both groups.
change of analgesia duration | first 24 hours postoperatively
  duration of analgesia was defined as the time from applying the block till the first intravenous morphine administration

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Fa Al-Rahamawy, MD, Study Chair — Professor of Anesthesia - Intensive Care Faculty of Medicine - Mansoura University; Hesham Ah Abdel Mohaiemn, MD, Study Director — Assistant Professor of Anesthesia - Intensive Care Faculty of Medicine - Mansoura University; Marwa Ib Abdo, MD, Principal Investigator — Lecturer of Anesthesia Intensive Care Faculty of Medicine - Mansoura University; Asmaa Ah Hossain, Ph.D, Principal Investigator — Residant in Anesthesia - Intensive Care Faculty of Medicine - Mansoura University
Locations (1):
- Marwa Ibrahim Mohamed Abdo, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal A, Batra RK, Chhabra A, Subramaniam R, Misra MC. The evaluation of efficacy and safety of paravertebral block for perioperative analgesia in patients undergoing laparoscopic cholecystectomy. Saudi J Anaesth. 2012 Oct-Dec;6(4):344-9. doi: 10.4103/1658-354X.105860. PMID 23493523
- [Background] Bisgaard T, Klarskov B, Rosenberg J, Kehlet H. Characteristics and prediction of early pain after laparoscopic cholecystectomy. Pain. 2001 Feb 15;90(3):261-269. doi: 10.1016/S0304-3959(00)00406-1. PMID 11207398
- [Background] Lau H, Brooks DC. Predictive factors for unanticipated admissions after ambulatory laparoscopic cholecystectomy. Arch Surg. 2001 Oct;136(10):1150-3. doi: 10.1001/archsurg.136.10.1150. PMID 11585507
- [Background] Salihoglu Z, Yildirim M, Demiroluk S, Kaya G, Karatas A, Ertem M, Aytac E. Evaluation of intravenous paracetamol administration on postoperative pain and recovery characteristics in patients undergoing laparoscopic cholecystectomy. Surg Laparosc Endosc Percutan Tech. 2009 Aug;19(4):321-3. doi: 10.1097/SLE.0b013e3181b13933. PMID 19692881
- [Background] Davies RG, Myles PS, Graham JM. A comparison of the analgesic efficacy and side-effects of paravertebral vs epidural blockade for thoracotomy--a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2006 Apr;96(4):418-26. doi: 10.1093/bja/ael020. Epub 2006 Feb 13. PMID 16476698
- [Background] Klein SM, Bergh A, Steele SM, Georgiade GS, Greengrass RA. Thoracic paravertebral block for breast surgery. Anesth Analg. 2000 Jun;90(6):1402-5. doi: 10.1097/00000539-200006000-00026. PMID 10825328
- [Background] Soni AK, Conacher ID, Waller DA, Hilton CJ. Video-assisted thoracoscopic placement of paravertebral catheters: a technique for postoperative analgesia for bilateral thoracoscopic surgery. Br J Anaesth. 1994 Apr;72(4):462-4. doi: 10.1093/bja/72.4.462. PMID 8155453
- [Background] Cheema SP, Ilsley D, Richardson J, Sabanathan S. A thermographic study of paravertebral analgesia. Anaesthesia. 1995 Feb;50(2):118-21. doi: 10.1111/j.1365-2044.1995.tb15092.x. PMID 7710020
- [Background] Kopacz DJ, Allen HW, Thompson GE. A comparison of epidural levobupivacaine 0.75% with racemic bupivacaine for lower abdominal surgery. Anesth Analg. 2000 Mar;90(3):642-8. doi: 10.1097/00000539-200003000-00026. PMID 10702451
- [Background] Bilgin M, Akcali Y, Oguzkaya F. Extrapleural regional versus systemic analgesia for relieving postthoracotomy pain: a clinical study of bupivacaine compared with metamizol. J Thorac Cardiovasc Surg. 2003 Nov;126(5):1580-3. doi: 10.1016/s0022-5223(03)00701-3. PMID 14666036
- [Background] Akhondzade R, Nesioonpour S, Gousheh M, Soltani F, Davarimoghadam M. The Effect of Magnesium Sulfate on Postoperative Pain in Upper Limb Surgeries by Supraclavicular Block Under Ultrasound Guidance. Anesth Pain Med. 2017 Jun 10;7(3):e14232. doi: 10.5812/aapm.14232. eCollection 2017 Jun. PMID 28924560
- [Background] Lee AR, Yi HW, Chung IS, Ko JS, Ahn HJ, Gwak MS, Choi DH, Choi SJ. Magnesium added to bupivacaine prolongs the duration of analgesia after interscalene nerve block. Can J Anaesth. 2012 Jan;59(1):21-7. doi: 10.1007/s12630-011-9604-5. Epub 2011 Oct 20. PMID 22012543
- [Background] Choyce A, Peng P. A systematic review of adjuncts for intravenous regional anesthesia for surgical procedures. Can J Anaesth. 2002 Jan;49(1):32-45. doi: 10.1007/BF03020416. PMID 11782326
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034